CLINICAL TRIAL: NCT03398304
Title: Defining the Temporal Changes in the Acute Phase Response During Graded Exercise: A Prospective Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jon Schoenecker, Associate Professor of Orthopaedic Surgery, Associate Professor of Pediatrics, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 171641
Record Dates: First submitted 2017-12-21; First posted 2018-01-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Phase Response
MeSH Terms: conditions — Acute-Phase Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graded Exercise (Experimental): Volunteers will participate in 3 study visits. The study visits will consist either of 20 minutes of walking, 20 minutes of running or 20 minutes of sitting. At the beginning of each study visit, prior to any exercise, a 4.5mL blood sample will be collected. The participant will then complete either 20 minutes of walking, running or sitting and will then have a 4.5mL blood draw taken from a new site.
  Interventions: Other: Graded Exercise
- Marathon Participation (Experimental): On the day of the marathon prior to start, the participant will be seated for 10 minutes prior to measuring their baseline heart rate. A 4.5 mL blood sample will be collected prior to initiation of exercise. Immediately after completion of the marathon, a 4.5 mL blood draw will be completed. Additional 4.5 mL blood draws will be taken at 1 and 2 days post-marathon to measure to length of time required to return to baseline coagulation, fibrinolysis, and inflammation following the prolonged, intense exercise.
  Interventions: Other: Marathon participation

INTERVENTIONS:
Other: Graded Exercise — Study arm 1 (Graded Exercise) participants will complete either 20 minutes of mild or moderate intensity at 2 different study visits. The third study visit will consist of 20 minutes of sitting.
  Arms: Graded Exercise
Other: Marathon participation — Study arm 2 (Marathon participation) participants will take part in a marathon. On the day of the marathon prior to start, the participant will be seated for 10 minutes prior to measuring their baseline heart rate. A 4.5 mL blood sample will be collected prior to initiation of exercise. Immediately after completion of the marathon, a 4.5 mL blood draw will be completed. Additional 4.5 mL blood draws will be taken at 1 and 2 days post-marathon to measure to length of time required to return to baseline coagulation, fibrinolysis, and inflammation following the prolonged, intense exercise.
  Arms: Marathon Participation

SUMMARY:
The purpose of this study is to detail the precise temporal changes in the APR that occur in response to exercise in order to determine the types of exercise that confer maximal reparative fibrinolysis. Published research and preliminary studies conducted in our lab suggest that different types of exercise will preferentially activate fibrinolysis over coagulation, thereby promoting improved global tissue health [8]. As such, measuring markers of the APR in healthy individuals 1) at rest, 2) walking (light intensity exercise), 3) running (moderate intensity exercise), and 4) following endurance running (a marathon) will allow us to establish a baseline for the temporal changes in the APR that avoid activation of the procoagulant survival phase while maximizing the repair phase.

Specific aims

1. To measure the acute phase response fibrinolysis, plasminogen consumption, and inflammatory profiles of healthy individuals before and after graded exercise (at rest, light intensity, medium intensity) and after prolonged exercise at medium intensity as defined by changes in fibrinolysis, plasminogen consumption, and inflammatory response.
2. To track the APR through modulated exercise in order to determine the type of exercise that enhances physiologic benefit and limits harm.

DETAILED DESCRIPTION:
Injury, ranging from a paper cut that barely splits the skin to a high-speed motor vehicle accident that rips through muscle and bone, causes a disruption of tissue compartments. This breach of compartments disposes tissue to four principle problems: 1) bleeding, 2) susceptibility to infection, 3) hypoxia, and 4) tissue dysfunction. The acute phase response (APR) is the physiologic system that resolves these four problems of injury. It is divided into two temporally distinct phases: survival and repair. The survival phase utilizes coagulation and inflammation to temporarily seal off breached compartments in order to stop bleeding and prevent the spread of infection. Once the life-threatening problems of hemorrhage and susceptibility to infection have been resolved, the body enters the repair phase, where it works to restore the disrupted blood supply and regenerate damaged tissue. These processes, coupled together, replace the temporary sealant and restore the injured tissue to its original form and function.

Plasmin is the key fibrinolytic protease that transitions the APR from survival to repair. Plasmin is traditionally known for its ability to degrade fibrin clots. Previous work has demonstrated that plasmin also activates many targets outside of fibrin degradation that are essential for musculoskeletal tissue healing. Plasmin initiates the repair of injured tissue by removing the temporary fibrin sealant required for hemostasis, which allows access for repair machinery to enter the site of injury. Subsequently, plasmin activates proteases that promote angiogenesis and cell differentiation to stimulate tissue regeneration. Without adequate plasmin activity, the body fails to transition from survival to repair and is unable to reconstitute the compartments damaged by injury.

All tissue injury activates the acute phase response. Exercise is a form of contained tissue injury that harnesses the beneficial effects of the acute phase response to build muscle and promote overall health. Given that the controlled injury of exercise minimizes compartment disruption, there is a limited need to mount a response to hemorrhage or containment of infection (survival). Exercise increases the metabolic requirement of muscle to the point that it outstrips the supply of oxygenated blood and results in sustained hypoxia. In response to hypoxia, plasmin stimulates angiogenesis and activates cells involved in tissue regeneration (repair). In exercise physiology, if major injury is avoided, the body thereby bypasses the survival phase and transitions into an early and prolonged repair phase.

Despite studies demonstrating alterations in the APR with exercise, the relationship between the intensity of exercise and the extent of APR activation is not yet well defined [8-10]. Our aim is to gain a better understanding of the precise changes in the APR in order to maximize the reparative potential of exercise. We hypothesize that moderate intensity exercise selectively enhances plasmin-mediated fibrinolysis (repair) without inducing the procoagulant arm of the APR (survival). Additionally, we propose that the systemic activation of fibrinolysis achieved in exercise promotes global tissue health at spatially distinct locations in addition to the site of initial tissue injury (hypoxic muscle). To evaluate this, we will define the precise temporal changes in the APR in healthy individuals participating in graded intensities of exercise (rest, light, and moderate). Through elucidation of the precise temporal activation of the APR as it relates to the intensity of exercise, it may allow future studies to develop an exercise regimen that harnesses the reparative potential of fibrinolysis while avoiding the potentially harmful activation of the procoagulant survival phase of the APR.

The purpose of this study is to detail the precise temporal changes in the APR that occur in response to exercise in order to determine the types of exercise that confer maximal reparative fibrinolysis. Published research and preliminary studies conducted in our lab suggest that different types of exercise will preferentially activate fibrinolysis over coagulation, thereby promoting improved global tissue health [8]. As such, measuring markers of the APR in healthy individuals 1) at rest, 2) walking (light intensity exercise), 3) running (moderate intensity exercise), and 4) following endurance running (a marathon) will allow us to establish a baseline for the temporal changes in the APR that avoid activation of the procoagulant survival phase while maximizing the repair phase.

Specific aims

1. To measure the acute phase response fibrinolysis, plasminogen consumption, and inflammatory profiles of healthy individuals before and after graded exercise (at rest, light intensity, medium intensity) and after prolonged exercise at medium intensity as defined by changes in fibrinolysis, plasminogen consumption, and inflammatory response.
2. To track the APR through modulated exercise in order to determine the type of exercise that enhances physiologic benefit and limits harm.

ELIGIBILITY:
Arm 1: 20-minute graded exercise Inclusion criteria

* Healthy individuals (male or female) aged 18-29
* Regular participation (at least 2 times per week) in moderate intensity exercise
* BMI between 18.5 and 30.0

Exclusion criteria

* Pre-existing health conditions or injuries that may limit the ability to safely participate in exercise
* Acute disease process such as an infection, broken bone, or asthma attack
* Chronic or recent use (within the last 10 days) of any anticoagulant medication or NSAID
* Pregnant women
* Recent inpatient admission within the last six months
* History of smoking or illicit drug use

Arm 2: Marathon participation Inclusion criteria

* Healthy individuals (male or female) aged 18-49
* In training to complete a marathon (individuals already planning on running a marathon and training accordingly for it)
* BMI between 18.5 and 30.0

Exclusion criteria

* Pre-existing health conditions or injuries that may limit the ability to safely participate in exercise
* Acute disease process such as an infection, broken bone, or asthma attack
* Chronic or recent use (within the last 10 days) of any anticoagulant medication or NSAID
* Pregnant women
* Recent inpatient admission within the last six months
* History of smoking or illicit drug use

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change of fibrinolysis (mg/ml) before graded exercise/marathon participation and after graded exercise/marathon participation (physiological parameter) | Baseline to post-exercise/marathon (within 3 hours of exercise/marathon completion)
  To measure the acute phase response fibrinolysis, plasminogen consumption, and inflammatory profiles of healthy individuals before and after graded exercise (at rest, light intensity, and medium intensity) and following endurance running, as defined by changes in fibrinolysis, plasminogen consumption, and inflammatory response.
Change of plasminogen (mg/ml) consumption before graded exercise/marathon participation and after graded exercise/marathon participation (physiological parameter) | Baseline to post-exercise/marathon (within 3 hours of exercise/marathon completion)
  To measure the acute phase response fibrinolysis, plasminogen consumption, and inflammatory profiles of healthy individuals before and after graded exercise (at rest, light intensity, and medium intensity) and following endurance running, as defined by changes in fibrinolysis, plasminogen consumption, and inflammatory response.
Change of inflammatory response (mg/ml) before graded exercise/marathon participation and after graded exercise/marathon participation (physiological parameter) | Baseline to post-exercise/marathon (within 3 hours of exercise/marathon completion)
  To measure the acute phase response fibrinolysis, plasminogen consumption, and inflammatory profiles of healthy individuals before and after graded exercise (at rest, light intensity, and medium intensity) and following endurance running, as defined by changes in fibrinolysis, plasminogen consumption, and inflammatory response.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Schoenecker, MD, PhD, Principal Investigator — Vanderbilt Orthopaedics
Locations (1):
- Vanderbilt Orthopaedics, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT03398304/ICF_001.pdf